CLINICAL TRIAL: NCT02977143
Title: Comparison of Positive End-expiratory Pressure-induced Increase in Central Venous Pressure and Stroke Volume Variation to Predict Fluid Responsiveness in Robot-assisted Laparoscopic Surgery: A Prospective Clinical Trial
Brief Title: Positive End-expiratory Pressure-induced Increase in Central Venous Pressure as a Predictor of Fluid Responsiveness in Robot-assisted Laparoscopic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Won Ho Kim, MD, Clinical Associate Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1609-101-793
Record Dates: First submitted 2016-11-27; First posted 2016-11-30 (Estimated); Last update posted 2018-04-03 (Actual); Status verified 2018-04

CONDITIONS: Prostatic Neoplasm; Urinary Bladder Neoplasm
Keywords: fluid responsiveness; central venous pressure; positive end-expiratory pressure; robot surgery
MeSH Terms: conditions — Prostatic Neoplasms; Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Fluid responsiveness test (Experimental): First, apply 10 cmH2O positive endexpiratory pressure (PEEP) and measure the increase in central venous pressure (CVP) as well as other preload indexes (central venous pressure, mean arterial pressure, stroke volume variation).
  Second, measure the increase in cardiac index after administration of volulyte 300 ml.
  If cardiac index increase more than 10%, fluid responsiveness is confirmed.
  Interventions: Procedure: Fluid loading of volulyte 300 ml

INTERVENTIONS:
Procedure: Fluid loading of volulyte 300 ml — Administration of volulyte 300 ml and measurement of increase in cardiac index

SUMMARY:
In urologic robotic surgery with steep Trendelenburg position, maintenance of cardiac preload and cardiac output is important for clinical prognosis. Previous studies reported the positive end-expiratory pressure (PEEP)-induced increase in central venous pressure (CVP) could be a accurate predictor of fluid responsiveness in cardiac surgical patients. The authors attempt to evaluate the predictability of PEEP-induced increase in CVP as well as stroke volume variation in urologic robotic surgery with Steep Trendelenburg position.

DETAILED DESCRIPTION:
In urologic robotic surgery with steep Trendelenburg position, maintenance of cardiac preload and cardiac output is important for clinical prognosis. As a preload index, the predictability of central venous pressure, pulse pressure variation and stroke volume variations may be impaired due to the impaired hemodynamics that result from the effect of increased abdominal pressure and decreased venous return. Previous studies reported the positive end-expiratory pressure (PEEP)-induced increase in central venous pressure (CVP) could be a accurate predictor of fluid responsiveness in cardiac surgical patients. Therefore, the authors attempt to evaluate the predictability of PEEP-induced increase in CVP as well as stroke volume variation in urologic robotic surgery with Steep Trendelenburg position.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient undergoing robot-assisted laparoscopic radical prostatectomy or cystectomy.
* American Society of Anesthesiologist Physical Status Classification of 1, 2 or 3.

Exclusion Criteria:

* Medical history of arrhythmia or new-onset arrhythmia after anesthesia induction.
* Valvular or ischemic heart disease or left ventricular ejection fraction less than 40%.
* Any significant pulmonary disease or history of chronic obstructive pulmonary disease
* End-stage renal disease or preoperative creatinine > 1.4 mg/dl

Min Age: 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
fluid responsiveness | 5 minutes after administration of 300 ml volulyte
  fluid responsiveness is determined when increase in cardiac index is more than 10%

SECONDARY OUTCOMES:
central venous pressure | one hour after the initiation of pneumoperitoneum
  T1: baseline measurement of central venous pressure with positive end-expiratory pressure of zero
cardiac index | one hour after the initiation of pneumoperitoneum
  T1: baseline measurement of cardiac index with positive end-expiratory pressure of zero
stroke volume variation | one hour after the initiation of pneumoperitoneum
  T1: baseline measurement of stroke volume variation with positive end-expiratory pressure of zero
abdominal pressure | one hour after the initiation of pneumoperitoneum
  T1: baseline measurement of abdominal pressure with positive end-expiratory pressure of zero
central venous pressure | 5 minutes after the application of positive end-expiratory pressure of 10 cmH2O
  T2: measurement of positive end-expiratory pressure-induce increase in central venous pressure
cardiac index | 5 minutes after the application of positive end-expiratory pressure of 10 cmH2O
  T2: measurement of cardiac index
stroke volume variation | 5 minutes after the application of positive end-expiratory pressure of 10 cmH2O
  T2: measurement of stroke volume variation
abdominal pressure | 5 minutes after the application of positive end-expiratory pressure of 10 cmH2O
  T2: measurement of abdominal pressure
central venous pressure | 5 minutes after removal of positive end-expiratory pressure
  T3: second baseline measurement of central venous pressure with positive end-expiratory pressure of zero
cardiac index | 5 minutes after removal of positive end-expiratory pressure
  T3: second baseline measurement of cardiac index with positive end-expiratory pressure of zero
stroke volume variation | 5 minutes after removal of positive end-expiratory pressure
  T3: second baseline measurement of stroke volume variation with positive end-expiratory pressure of zero
abdominal pressure | 5 minutes after removal of positive end-expiratory pressure
  T3: second baseline measurement of abdominal pressure with positive end-expiratory pressure of zero
central venous pressure | T4: 5 minutes after administration of volulyte 300 ml
  measurement of central venous pressure after fluid administration
cardiac index | T4: 5 minutes after administration of volulyte 300 ml
  measurement of cardiac index after fluid administration
stroke volume variation | T4: 5 minutes after administration of volulyte 300 ml
  measurement of stroke volume variation after fluid administration
abdominal pressure | T4: 5 minutes after administration of volulyte 300 ml
  measurement of abdominal pressure after fluid administration
arterial oxygen partial pressure (mmHg) | 5 minutes after anesthesia induction
  arterial blood gas analysis
arterial carbon dioxide partial pressure (mmHg) | 5 minutes after anesthesia induction
  arterial blood gas analysis
arterial oxygen partial pressure (mmHg) | 1 minutes after the application of positive end-expiratory pressure of 10 cmH2O
  arterial blood gas analysis
arterial carbon dioxide partial pressure (mmHg) | 1 minutes after the application of positive end-expiratory pressure of 10 cmH2O
  arterial blood gas analysis
arterial oxygen partial pressure (mmHg) | 1 minutes after the start of skin closure
  arterial blood gas analysis
arterial carbon dioxide partial pressure (mmHg) | 1 minutes after the start of skin closure
  arterial blood gas analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No